CLINICAL TRIAL: NCT06814847
Title: Interpretation of Uroflowmetry Samples from Pediatric Patients by Clinicians and Introduction to Artificial Intelligence, and Interpretation of the Samples by Artificial Intelligence
Brief Title: Artificial Intelligence-Based Analysis of Uroflowmetry Patterns in Children: a Machine Learning Perspective
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: MAR.UAD.0019
Record Dates: First submitted 2025-02-03; First posted 2025-02-07 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Voiding Dysfunction; Voiding Disorders; Machine Learning
Keywords: Uroflowmetry voiding patterns; Interpretation differences; Machine learning; Artificial intelligence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Uroflowmetry is the one of the most commonly used non-invasive test for evaluating children with lower urinary tract symptoms (LUTS). However, studies have highlighted a weak agreement among experts in interpreting uroflowmetry patterns. This study aims to assess the impact of machine learning models, which have become increasingly prevalent in medicine, on the interpretation of uroflowmetry patterns.

DETAILED DESCRIPTION:
The study included uroflowmetry tests of children aged 4-17 years who were referred to our clinic with lower urinary tract symptoms. Uroflowmetry patterns were independently interpreted by three pediatric urology experts. Discrepancies in interpretations were jointly re-evaluated by the three observers, and a consensus was reached. Voiding volume, voiding duration, and urine flow rates at 0.5-second intervals were converted into numerical data for analysis. Eighty percent of the dataset was used as training data for machine learning, while there maining 20% was reserved for testing. A total of five different machine learning models were employed for classification: Decision Tree, Random Forest, CatBoost, XGBoost, and LightGBM. The models that most accurately identified each uroflowmetry pattern were determined.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 4 and 17 years with LUTS
* Urinate more than 50% of the expected bladder capacity on UF

Exclusion Criteria:

* Patients who were unable to cooperate with the voiding command
* Had neurological disorders
* Urinate less than 50% of the expected bladder capacity on UF
* Under 4 years of age, and were over 18 years of age

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children aged 4-17
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Performance of Machine Learning Models in Evaluating Voiding Patterns | From October 2024 to January 2025
  5 different machine learning models were used. Accuracy rates were determined for each model.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University School of Medicine, Urology Department, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Arslan F, Algorabi O, Ozkan OC, Turkan YS, Ersin Namli, Genc YE, Sekerci CA, Yucel S, Cam K, Tarcan T. Artificial Intelligence-Based Analysis of Uroflowmetry Patterns in Children: A Machine Learning Perspective. Neurourol Urodyn. 2025 Nov;44(8):1575-1582. doi: 10.1002/nau.70139. Epub 2025 Sep 4. PMID 40908659